CLINICAL TRIAL: NCT00001059
Title: Comparison Study of Liposomal Doxorubicin With or Without Bleomycin and Vincristine for the Treatment of Advanced AIDS-Associated Kaposi's Sarcoma
Brief Title: Comparison of Liposomal Doxorubicin Used Alone or in Combination With Bleomycin Plus Vincristine in the Treatment of Kaposi's Sarcoma in Patients With AIDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Sequus Pharmaceuticals (Industry); Amgen (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 286; 11262 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Vincristine; Sarcoma, Kaposi; Liposomes; Doxorubicin; Drug Therapy, Combination; Granulocyte Colony-Stimulating Factor; Acquired Immunodeficiency Syndrome; Bleomycin; Drug Carriers
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Doxorubicin; Liposomes; Filgrastim; Bleomycin; Vincristine

INTERVENTIONS:
Drug: Doxorubicin hydrochloride (liposomal)
Drug: Filgrastim
Drug: Bleomycin sulfate
Drug: Vincristine sulfate

SUMMARY:
To evaluate the safety and efficacy of liposomal doxorubicin hydrochloride ( DOX-SL ) alone or in combination with bleomycin and vincristine in the long-term treatment of AIDS-related Kaposi's sarcoma. To determine whether the 3-drug combination enhances progression-free survival and quality of life.

Liposomal formulations of chemotherapeutic agents increase drug accumulation in tumors, which permits disease palliation at relatively low doses and thus decreases some of the dose-limiting toxicity. Multi-agent therapy is considered to be more effective than single-agent therapy; therefore, DOX-SL will be combined with bleomycin and vincristine.

DETAILED DESCRIPTION:
Liposomal formulations of chemotherapeutic agents increase drug accumulation in tumors, which permits disease palliation at relatively low doses and thus decreases some of the dose-limiting toxicity. Multi-agent therapy is considered to be more effective than single-agent therapy; therefore, DOX-SL will be combined with bleomycin and vincristine.

Patients are randomized to receive intravenous DOX-SL alone or in combination with vincristine/bleomycin every 2 weeks. Filgrastim ( granulocyte colony-stimulating factor; G-CSF ) may be given as needed for neutropenia.

AS PER AMENDMENT 11/7/96: Based on interim review data, it is recommended that subjects receiving DOX-SL plus vincristine/bleomycin have vincristine/bleomycin discontinued and receive DOX-SL alone unless, in the opinion of the treating physician, they are benefitting from the DOX-SL plus vincristine/bleomycin regimen.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* G-CSF.
* Licensed or Treatment IND-approved antiretrovirals ( AZT, ddI, ddC, d4T ).
* PCP prophylaxis (required if CD4 count < 200 cells/mm3).
* Chemoprophylaxis or maintenance for bacterial infections, candidiasis, MAC, and herpes simplex.
* Up to 14 days of metronidazole.
* Recombinant erythropoietin.

Patients must have:

* Documented HIV infection.
* Advanced stage Kaposi's sarcoma.
* No active acute opportunistic infection.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Significant pulmonary insufficiency (unless due to pulmonary KS).
* Significant cardiac insufficiency.
* Other active malignancies except for basal or squamous cell carcinoma of the skin or in situ cervical cancer.
* Grade 2 or worse peripheral neuropathy.
* Altered mental status that prevents informed consent.
* Active Mycobacterium tuberculosis.
* Hypersensitivity or allergic reaction to any study drugs or E. coli-derived medications such as filgrastim (G-CSF).

Concurrent Medication:

Excluded:

* GM-CSF.
* Drugs associated with peripheral neuropathy (other than approved antiretrovirals and vincristine).
* Multi-drug therapy for active Mycobacterium tuberculosis (although isoniazid and pyridoxine is allowed as treatment for a positive PPD, with permission of study chair).

Concurrent Treatment:

Excluded:

* Radiation therapy to study marker lesions.

Patients with the following prior condition are excluded:

* Neuropsychiatric history.

Prior Medication:

Excluded:

* Any anti-KS therapy within 21 days prior to study entry.
* Prior systemic therapy with any anthracycline (including liposomal anthracyclines), vincristine, or bleomycin.
* Any investigational drug (other than those available through Treatment IND and used for FDA-sanctioned purposes) within 14 days prior to study entry.

PER AMENDMENT 11/29/95:

* No more than 2 cycles of any systemic chemotherapy for Kaposi's sarcoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Study Completion 1998-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitsuyasu R, Study Chair; Krown S, Study Chair; Von Roenn JH, Study Chair
Locations (17):
- United States (17):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Ucsf Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Queens Med. Ctr., Honolulu, Hawaii
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Memorial Sloan-Kettering Cancer Ctr., New York, New York

REFERENCES:
- [Background] Mitsuyasu R, et al. Comparison study of liposomal doxorubicin (DOX) alone or with bleomycin and vincristine (DBV) for treatment of advanced AIDS-associated Kaposi's sarcoma (AIDS-KS): AIDS Clinical Trial Group (ACTG) protocol 286 (meeting abstract). Proc Annu Meet Am Soc Clin Oncol. 1997;16:A191